CLINICAL TRIAL: NCT03052387
Title: Assessment of Vertical Bone Augmentation Using Autogenous Onlay Versus Inlay Grafting Techniques With Simultaneous Implant Placement in the Anterior Maxillary Area on Patient's Esthetic Satisfaction : A Randomized Clinical Trial
Brief Title: Vertical Augmentation Using Onlay Versus Inlay Autogenous Graft With Simultaneous Implant Placement.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Ahmed Hassan, Dentist at National research centre, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CairoAMI-CG
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): * Crestal pyramidal flap will be done with 2 releasing incisions for adequate exposure.
  * Buccal& palatal full reflection for adequate exposure and to avoid the interference between the onlay graft and the residual bone.
  * Decortication of the bone bed to increase the blood supply to the onlay graft.
  * The block graft harvested from the chin is placed crestal to the residual ridge and stabilized in place using dental implant immediately.
  * Periosteal incisions are usually needed to allow tension free sutures.
  * Vicryl 3/0 sutures for closer.
  * augmentin 1g twice daily for 5 days.
  * catflam 50g twice daily for 3 days
  Interventions: Other: assigned intervention
- Comparator (Active Comparator): * Crestal incision with labial flap reflected leaving the palatal tissues without elevation.
  * Marking of the 3 bony cuts ( 2 vertical cuts & 1 horizontal cut ) using fine fissure bur in the form of perforations along the cuts position.
  * Drilling of pilot drill and first drill only.
  * 3 full thickness cuts will be performed (2 vertical stop cuts will be made by using the tungsten carbide disc at the distal ends of the horizontal bony cut on the facial surface of alveolar ridge.
  * splitting osteotomes are used and mallet to complete the splitting of the bony segment.
  * After bony separation the rectangular bony segment (transport segment) will be mobilized occlusally and pedicled on the palatal mucoperiosteum.
  * The autogenous block graft harvested from the chin area is placed in the space gained under the mobile bony segment.
  * Drilling through the bony segment and the block graft.
  * Immediate implant placement
  chin graft block dental implants
  Interventions: Other: assigned intervention

INTERVENTIONS:
Other: assigned intervention — * Local anesthesia with vasoconstrictor(V.C) used for hemostasis.
  chin block graft
  * Scrubbing and draping of the patient will be carried out in a standard fashion using betadine surgical scrub.
  * The donor site is usually the chin area, its approached using local anesthesia with VC at symphysis region.
  * Low vestibular incision exposing the symphysis area to the inferior border of the mandible.
  * Using fissure bur to harvest the graft for the defect.
  * Closure using vicryl 3-O sutures.

SUMMARY:
Using autogenous Chin block for vertical augmentation with simultaneous implant placement at anterior maxilla region comparing between the Onlay and Inlay grafting techniques.

DETAILED DESCRIPTION:
to study the vertical augmentation with simultaneous implant placement at anterior maxillary region.

* P: Patient requires implant at anterior maxillary ridge with vertical deficiency.
* I:Inlay Sandwich Technique with immediate implant placement.
* C:Onlay autogenous graft immediate implant placement.
* O:Outcome name Measuring device Measuring unit

Primary outcome: Vertical bone gain CBCT Millimeter

-Secondary outcome(a): Crestal bone loss CBCT Millimeter

ELIGIBILITY:
Inclusion Criteria:

* * Patients with partially edentulous anterior maxillary ridges.

  * Patients were free from any systemic disease that interferes with bone healing.
  * Absence of local pathosis at anterior maxillary area.
  * No history of any grafting procedure at the designated edentulous ridge.

The edentulous ridge vertical dimension was less than 10 mm measured from the alveolar crest to the nasal floor (i.e.ridge had vertical inadequacy) with normal horizontal alveolar dimension or patient with Increased Inter-Arch Space.

Exclusion Criteria:

* * Patient with fully dentulous maxilla.

  * Pregnant females.
  * Presence of bad habits (severe bruxism, clenching).
  * Systemic diseases that may interfere with bone healing.e.g. uncontrolled Diabetes.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
vertical Bone gain | 6 months
  * The nasal floor will be used as a fixed reference by adjusting the cross sectional long axis in the center of the area of interest and bisecting it (showing the buccolingual dimension).
  * All the patients will wear the radiographic dentures with radiopaque material (barium sulphate mixed with acrylic powder) filling the teeth at the area of interest to ensure that the calculations were taken at the same region.
  * On the cross sectional view of CBCT and at each proposed implant site, a line will be drawn starting from the crest of the ridge till the nasal floor. The height will be recorded preoperatively, immediately (1 week) and 6 months postoperatively.the difference between them in millimeters will be recorded.

SECONDARY OUTCOMES:
crestal bone loss | 6 months
  crestal bone loss around the implant will be measured in millimeter after 6 months

IPD SHARING:
Plan to Share IPD: No
assessment of vertical ridge augmentation using autogenous Onlay versus Inlay Bone Grafting techniques in the anterior maxilla.